CLINICAL TRIAL: NCT03708497
Title: The Effect of Carbetocin Versus Oral Tranexamic Acid Plus, Buccal Misoprostol on Blood Loss After Vaginal Delivery: a Randomized Controlled Trial
Brief Title: Carbetocin Versus Oral Tranexamic Acid Plus, Buccal Misoprostol on Blood Loss After Vaginal Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aswan University Hospital (Other)
Responsible Party: Principal Investigator, hany farouk, lecturer, Aswan University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: aswu/293/9/18
Record Dates: First submitted 2018-10-13; First posted 2018-10-17 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-08

CONDITIONS: Postpartum Hemorrhage
Keywords: carbetocin; tranexamic acid; postpartum hemorrhage; buccal misoprostol
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — carbetocin; Tranexamic Acid; Misoprostol

STUDY DESIGN:
Intervention Model Description: women were allocated to one of the three study groups: group I (carbetocin group) received 100 mc carbetocin IV after delivery of the baby, group II (misoprostol group) received 600 mg buccal misoprostol after delivery of the baby, and group III (TA plus misoprostol group) received 1000mg oral TA at the end of the first stage of labor plus 600 mg buccal misoprostol after delivery of the baby. A buccal route, in which the tablets are placed in the cheek for 30 min after which any remnants are swallowed
Masking Description: open label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- carbetocin (Active Comparator): Carbetocin 100 microgram will be applied intravenously in a short infusion over about a minute
  Interventions: Drug: carbetocin
- Tranexamic acid plus misoprostol (Experimental): 1000mg oral TA at the end of the first stage of labor plus 600 mg buccal misoprostol after delivery of the baby. A buccal route, in which the tablets are placed in the cheek for 30 min after which any remnants are swallowed.
  Interventions: Drug: Tranexamic acid plus misoprostol
- misoprostol (Active Comparator): 600 mg buccal misoprostol after delivery of the baby. A buccal route, in which the tablets are placed in the cheek for 30 min after which any remnants are swallowed.
  Interventions: Drug: misoprostol

INTERVENTIONS:
Drug: carbetocin — Carbetocin 100 microgram will be applied intravenously in a short infusion over about a minute
  Other Names: Active Comparator
  Arms: carbetocin
Drug: Tranexamic acid plus misoprostol — 1000mg oral TA at the end of the first stage of labor plus 600 mg buccal misoprostol after delivery of the baby. A buccal route, in which the tablets are placed in the cheek for 30 min after which any remnants are swallowed.
  Other Names: active comparator
  Arms: Tranexamic acid plus misoprostol
Drug: misoprostol — 600 mg buccal misoprostol after delivery of the baby. A buccal route, in which the tablets are placed in the cheek for 30 min after which any remnants are swallowed.
  Other Names: active comparator
  Arms: misoprostol

SUMMARY:
Excessive bleeding at or after childbirth accounts for about half of all the post-partum maternal deaths in developing countries and is the single most important cause of maternal mortality worldwide. Post-partum hemorrhage (PPH) is the major contributor to maternal mortality worldwide representing at least 25% of the maternal deaths annually. Prevention of PPH has become a global aim to reduce maternal mortality. Uterine atony is the main cause of PPH; therefore, active management of the third stage of labor has emerged as a most actual tool in its prevention. The previous study in Egypt recorded that 88% of deaths from PPH occur within 4 hours of delivery. Tranexamic acid (TA) is an antifibrinolytic agent that blocks the lysine-binding site of plasminogen to fibrin. Misoprostol is effective when given orally, buccal, sublingually, vaginally, or rectally, so it might be used by traditional birth attendants, or self-administered, in cases of home-births occurred without the attendance of health personnel or where women are at most risk for occurrence of severe PPH. So, the current study aims to evaluate the effect of prophylactic oral TA plus buccal misoprostol in the prevention of primary PPH after routine active management of the third stage of labor in women at low risk for uterine atony in comparison with carbetocin and buccal misoprostol alone.

DETAILED DESCRIPTION:
All women admitted to the reception unit for vaginal delivery were invited to participate in the study. The investigators included women aged (20-35 years) with a singleton pregnancy in a cephalic presentation between 38 and 42 weeks gestation. The participated women have entered the screening phase of the study. This phase included history taking (age, parity, and gestational age) with measurement of weight, temperature, and initial hemoglobin level. The investigators excluded women with medical disorders such as cardiac, hepatic, renal, neurologic disorders thromboembolic disease, blood disorders, diabetes, gestational hypertension, and pre-eclampsia. Women at risk for PPH as grand multipara (parity >5), multiple pregnancies, polyhydramnios, fetal macrosomia, antepartum hemorrhage, prolonged, and obstructed labor were also excluded. Moreover, we excluded women with a scarred uterus or previous instrumental delivery and those suffering from hypersensitivity to TA. women were allocated to one of the three study groups: group I (carbetocin group) received 100 mc carbetocin IV after delivery of the baby, group II (misoprostol group) received 600 mg buccal misoprostol after delivery of the baby, and group III (TA plus misoprostol group) received 1000mg oral TA at the end of the first stage of labor plus 600 mg buccal misoprostol after delivery of the baby. A buccal route, in which the tablets are placed in the cheek for 30 min after which any remnants are swallowed.

ELIGIBILITY:
Inclusion Criteria:

* All women admitted to the reception unit for vaginal delivery
* women aged (20-35 years) with a singleton pregnancy in a cephalic presentation between 38 and 42 weeks gestation.

Exclusion Criteria:

* medical disorders such as cardiac, hepatic, renal, neurologic disorders thromboembolic disease, blood disorders, diabetes, gestational hypertension, and pre-eclampsia.

-Women at risk for PPH as grand multipara (parity >5), multiple pregnancies, polyhydramnios, fetal macrosomia, antepartum hemorrhage, prolonged, and obstructed labor were also excluded.-

* Moreover, we excluded women with a scarred uterus or previous instrumental delivery and those suffering from hypersensitivity to TA.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — All women admitted to the reception unit for vaginal delivery were invited to participate in the study
Enrollment: 360 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
difference in the mean blood loss at 4 h postpartum between the three groups | 4 hours post delivery
  measure blood loss by direct and gravimetric methods

SECONDARY OUTCOMES:
difference in hemoglobin level | 24 hours postdelivery
  hemoglobin level pre delivery and 24 hours post delivery
the need for additional uterotonics | ist 24 hours postoperative
  the need of additional oxytocin or misoprostol

CONTACTS AND LOCATIONS:
Overall Officials: hany f sallam, md, Principal Investigator — Aswan University Hospital
Locations (2):
- Egypt (2):
  - Aswan University, Aswān
  - AswanUH, Aswān

IPD SHARING:
Plan to Share IPD: No